CLINICAL TRIAL: NCT02814916
Title: A Phase 3, Multicenter, Open-Label, Randomized, Comparator Controlled Trial of the Safety and Efficacy of Dalbavancin Versus Active Comparator in Pediatric Subjects With Acute Bacterial Skin and Skin Structure Infections
Brief Title: Dalbavancin for the Treatment of Acute Bacterial Skin and Skin Structure Infections in Children, Known or Suspected to be Caused by Susceptible Gram-positive Organisms, Including MRSA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DUR001-306; 2014-005281-30 (EudraCT Number)
Record Dates: First submitted 2016-06-08; First posted 2016-06-28 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Methicillin-Resistant Staphylococcus Aureus; Bacterial Infections; Staphylococcal Skin Infections
Keywords: Acute Bacterial Skin and Skin Structure Infection (ABSSSI)
MeSH Terms: conditions — Bacterial Infections; Staphylococcal Skin Infections | interventions — dalbavancin; Vancomycin; Oxacillin; Floxacillin; Cefadroxil; Clindamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dalbavancin single-dose (Experimental): Participants received dalbavancin administered intravenously as follows: birth to < 3 months old and 3 months to < 6 years old: 22.5 mg/kg (maximum 1500 mg) on Day 1; ≥6 years to 17 years old (inclusive): 18 mg/kg (maximum 1500 mg) on Day 1. Participants aged birth to < 3 months were not randomized; all received dalbavancin single-dose.
  Interventions: Drug: Dalbavancin
- Dalbavancin two-dose (Experimental): Participants received dalbavancin administered intravenously as follows: 3 months to < 6 years old: 15 mg/kg (maximum 1000 mg) on Day 1, and 7.5 mg/kg (maximum 500 mg) on Day 8; ≥6 years to 17 years old (inclusive): 12 mg/kg (maximum 1000 mg) on Day 1, and 6 mg/kg (maximum 500 mg) on Day 8.
  Interventions: Drug: Dalbavancin
- Comparator (Active Comparator): Participants 3 mos to < 6 yrs old and ≥6 yrs to 17 yrs old received a 10-14 day course of either vancomycin 10 to 15 mg/kg/dose, not to exceed a 4000 mg total daily dose; or oxacillin 30 mg/kg/dose, infused over 60 (± 10) mins every 6 (± 1) hrs; or flucloxacillin 50 mg/kg/dose, infused over 60 (± 10) mins every 6 (± 1) hrs, not to exceed a 2000 mg total daily dose. Vancomycin was to be taken for methicillin-resistant Gram-positive infections. Based on local practice patterns/approvals for clinical use in the pediatric population, oxacillin or flucloxacillin were supplied as an IV comparator. At investigator's discretion, after 72 hrs of IV therapy, those on oxacillin or flucloxacillin could switch to oral cefadroxil (dose for infants/children: 15 mg/kg/dose every 12 hrs, max 2 g/day; dose for adolescents: 500-1000 mg every 12 hrs), and if infection with methicillin-resistant S. aureus was confirmed, those on vancomycin were allowed to switch to oral clindamycin 10 mg/kg every 8 hrs.
  Interventions: Drug: Vancomycin; Drug: Oxacillin; Drug: Flucloxacillin; Drug: Cefadroxil; Drug: Clindamycin

INTERVENTIONS:
Drug: Dalbavancin — Dalbavancin was administered intravenously over 30 (± 5) minutes.
  Other Names: Xydalba
  Arms: Dalbavancin single-dose; Dalbavancin two-dose
Drug: Vancomycin — Vancomycin was administered intravenously over 60 (± 10) minutes every 6 (± 1) hours.
  Arms: Comparator
Drug: Oxacillin — Oxacillin was administered intravenously over 60 (± 10) minutes every 6 (± 1) hours.
  Arms: Comparator
Drug: Flucloxacillin — Flucloxacillin was administered intravenously over 60 (± 10) minutes every 6 (± 1) hours.
  Arms: Comparator
Drug: Cefadroxil — Cefadroxil was administered orally every 12 hours.
  Arms: Comparator
Drug: Clindamycin — Clindamycin was administered orally every 8 hours.
  Arms: Comparator

SUMMARY:
To determine the safety and descriptive efficacy of dalbavancin for the treatment of acute bacterial skin and skin structure infections in children, aged birth to 17 years (inclusive), known or suspected to be caused by susceptible Gram-positive organisms, including methicillin-resistant strains of Staphylococcus aureus.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients birth to 17 years (inclusive)
* A clinical picture compatible with Acute Bacterial Skin and Skin Structure Infections (ABSSSI) suspected or confirmed to be caused by Gram-positive bacteria, including Methicillin-resistant Staphylococcus aureus (MRSA).
* In addition to local signs of ABSSSI, the patient has at least one of the following:
* Fever, defined as body temperature ≥ 38.4°C (101.2°F) taken orally, ≥ 38.7°C (101.6°F) tympanically, or ≥ 39°C (102.2°F) rectally (core temperature) OR
* Leukocytosis (WBC > 10,000 mm3) or leukopenia (WBC < 2,000 mm3) or left shift of >10% band neutrophils
* Infection either involving deeper soft tissue or requiring significant surgical intervention
* Major cutaneous abscess characterized as a collection of pus within the dermis or deeper that is accompanied by erythema, edema and/or induration which i. requires surgical incision and drainage, and ii. is associated with cellulitis such that the total affected area involves at least 35 cm2 of erythema, or total affected area of erythema is at least BSA (m2) x 43.0 (cm2/m2), OR iii. alternatively, involves the central face and is associated with an area of erythema of at least 15 cm2 b. Surgical site or traumatic wound infection characterized by purulent drainage with surrounding erythema, edema and/or induration which occurred within 30 days after the trauma or surgery and is associated with cellulitis such that: i. the total affected area involves at least 35 cm2 of erythema, or total affected area of erythema is at least BSA (m2) x 43.0 (cm2/m2), OR ii. alternatively, involves the central face and is associated with an affected area of at least 15 cm2 c. Cellulitis, defined as a diffuse skin infection characterized by spreading areas of erythema, edema and/or induration and: i. is associated with erythema that involves at least 35 cm2 of surface area, or surface area of erythema is at least BSA (m2) x 43.0 (cm2/m2), OR ii. alternatively, cellulitis of the central face that is associated with an affected area of at least 15 cm2 5. In addition to the requirement for erythema, all patients are required to have at least two (2) of the following signs of ABSSSI: a. Purulent drainage/discharge b. Fluctuance c. Heat/localized warmth d. Tenderness to palpation e. Swelling/induration

  * In patients age birth to < 3 months, each patient must meet the following inclusion criteria to be enrolled in this study.

    1. Male or female patients from birth to < 3 months of age, including pre-term neonates (gestational age ≥ 32 weeks)
    2. A clinical picture compatible with an ABSSSI suspected or confirmed to be caused by Gram-positive bacteria, including MRSA.

       OR

       Suspected or confirmed sepsis including any of the following clinical criteria:
       1. Hypothermia (<36°C) OR fever (>38.5°C)
       2. Bradycardia OR tachycardia OR rhythm instability
       3. Hypotension OR mottled skin OR impaired peripheral perfusion
       4. Petechial rash
       5. New onset or worsening of apnea episodes OR tachypnea episodes OR increased oxygen requirements OR requirement for ventilation support
       6. Feeding intolerance OR poor sucking OR abdominal distension
       7. Irritability
       8. Lethargy
       9. Hypotonia
    3. In addition, patients must meet at least one of the following laboratory criteria:

       a. White blood cell count ≤4.0 × 10^9/L OR ≥20.0 × 10^9/L b, Immature to total neutrophil ratio >0.2 c. Platelet count ≤100 × 10^9/L d. C-reactive protein (CRP) >15 mg/L OR procalcitonin ≥ 2 ng/mL e. Hyperglycemia OR Hypoglycemia f. Metabolic acidosis
    4. Infections must be of sufficient severity to merit hospitalization and parenteral antibiotic therapy. These infections may include:

       1. Cutaneous or subcutaneous abscess
       2. Surgical site or traumatic wound infection
       3. Cellulitis, Erysipelas
       4. Omphalitis
       5. Impetigo and bullous impetigo
       6. Pustular folliculitis
       7. Scarlet fever
       8. Staphylococcal scalded skin syndrome
       9. Streptococcal toxic shock syndrome
       10. Erythematous based-erosion
       11. Other infections originating in the skin or subcutaneous tissue and associated with signs and symptoms of sepsis as defined in Inclusion Criterion 2.
    5. Patients must be expected to survive with appropriate antibiotic therapy and appropriate supportive care throughout the study.

Exclusion Criteria:

1. Patients age 3 months to 17 years: Clinically significant renal impairment, defined as calculated creatinine clearance of less than 30 mL/min. (calculated by the Schwartz "bedside" formula). Patients birth to < 3 months of age: Moderate or severe renal impairment defined as serum creatinine ≥ 2 times the upper limit of normal (× ULN) for age OR urine output < 0.5 mL/kg/h (measured over at least 8 hours prior to dosing) OR requirement for dialysis.
2. Clinically significant hepatic impairment, defined as serum bilirubin or alkaline phosphatase greater than 2 times the upper limits of normal (ULN) for age, and/or serum aspartate aminotransferase (AST) or alanine transaminase (ALT) greater than 3 times the upper limits of normal (ULN) for age.
3. Treatment with an investigational drug within 30 days preceding the first dose of study medication.
4. Patients with sustained shock defined as systolic blood pressure < 90 mm Hg in children ≥ 10 years old, < 70 mm Hg + [2 x age in years] in children 1 to <10 years, or < 70 mmHg in infants 3 to <12 months old for more than 2 hours despite adequate fluid resuscitation, with evidence of hypoperfusion or need for sympathomimetic agents to maintain blood pressure.
5. More than 24 hours of any systemic antibacterial therapy within 96 hours before randomization. EXCEPTION: Microbiological or clinical treatment failure with a systemic antibiotic other than IV study drug that was administered for at least 48 hours. Failure must be confirmed by either a microbiological laboratory report or documented worsening clinical signs or symptoms.
6. Infection due to an organism known prior to study entry to be resistant to dalbavancin (dalbavancin minimum inhibitory concentration (MIC) greater than 0.25 ug/mL) or vancomycin (vancomycin minimum inhibitory concentration (MIC) greater than 2 ug/mL).
7. Patients with necrotizing fasciitis, or deep-seated infections that would require > 2 weeks of antibiotics (e.g., endocarditis, osteomyelitis or septic arthritis).
8. Infections caused exclusively by Gram-negative bacteria (without Gram-positive bacteria present) and infections caused by fungi, whether alone or in combination with a bacterial pathogen.
9. Venous catheter entry site infection.
10. Infections involving diabetic foot ulceration, perirectal abscess or a decubitus ulcer.
11. Patient with an infected device, even if the device is removed. Examples include infection of: prosthetic cardiac valve, vascular graft, a pacemaker battery pack, joint prosthesis, implantable pacemaker or defibrillator, intraaortic balloon pump, left ventricular assist device, or a neurosurgical device such as a ventricular peritoneal shunt, intra-cranial pressure monitor, or epidural catheter.
12. Gram-negative bacteremia, even in the presence of Gram-positive infection or Gram-positive bacteremia. Note: If a Gram-negative bacteremia develops during the study, or is subsequently found to have been present at Baseline, the patient should be removed from study treatment and receive appropriate antibiotic(s) to treat the Gram-negative bacteremia.
13. Patients whose skin infection is the result of having sustained full or partial thickness burns.
14. Patients age 3 months to 17 years, with uncomplicated skin infections such as superficial/simple cellulitis/erysipelas, impetiginous lesion, furuncle, or simple abscess that only requires surgical drainage for cure. Patients birth to < 3 months of age may be enrolled if they have uncomplicated skin infections of sufficient severity to require hospitalization and parenteral antibiotic therapy.
15. Patients age 3 months to 17 years: Concomitant condition requiring any antibiotic therapy that would interfere with the assessment of study drug for the condition under study.
16. Sickle cell anemia
17. Cystic fibrosis
18. Anticipated need of antibiotic therapy for longer than 14 days.
19. Patients who are placed in a hyperbaric chamber as adjunctive therapy for the ABSSSI.
20. More than 2 surgical interventions (defined as procedures conducted under sterile technique and typically unable to be performed at the bedside) for the skin infection, or patients who are expected to require more than 2 such interventions.
21. Medical conditions in which chronic inflammation may preclude assessment of clinical response to therapy even after successful treatment (e.g., chronic stasis dermatitis of the lower extremity).
22. Immunosuppression/immune deficiency, including hematologic malignancy, recent bone marrow transplant (in post-transplant hospital stay), absolute neutrophil count < 500 cells/mm3, receiving immunosuppressant drugs after organ transplantation, receiving oral steroids ≥ 20 mg prednisolone per day (or equivalent) for > 14 days prior to enrollment, and known or suspected human immunodeficiency virus (HIV) infected patients with a CD4 cell count< 200 cells/mm3 or with a past or current acquired immunodeficiency syndrome (AIDS)-defining condition and unknown CD4 count.
23. Known or suspected hypersensitivity to glycopeptide antibiotics, betalactam agents, aztreonam, or cephalosporins.
24. Patients with a rapidly fatal illness, who are not expected to survive for 3 months.
25. Positive urine (or serum) pregnancy test at screening (post-menarchal females only) or after admission (prior to dosing).
26. Pregnant or nursing females; sexually active females of childbearing potential who are unwilling or unable to use adequate contraceptive precautions. Female patients to have pregnancy testing are those who are at least 10 years old with menarche and/or thelarche (beginning of breast development).

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 199 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (84):
- United States (15):
  - University of South Alabama /ID# 237446, Mobile, Alabama
  - Valleywise Health Medical Center /ID# 234343, Phoenix, Arizona
  - Southbay Pharma Research /ID# 235700, La Palma, California
  - University of California, Los Angeles /ID# 237533, Los Angeles, California
  - Duplicate_Children's Hospital Colorado /ID# 237622, Aurora, Colorado
  - Global Research Holdings LLC /ID# 235747, Panama City, Florida
  - Tampa General Hospital /ID# 237061, Tampa, Florida
  - Children's Healthcare of Atlanta - Ferry Rd /ID# 237003, Atlanta, Georgia
  - University of Maryland Medical Center /ID# 234353, Baltimore, Maryland
  - Duplicate_Children's Mercy Hospital and Clinics /ID# 237800, Kansas City, Missouri
  - Robert Wood Johnson Univ Hosp /ID# 237862, New Brunswick, New Jersey
  - NYU School of Medicine /ID# 236783, New York, New York
  - SUNY Upstate Medical University /ID# 236831, Syracuse, New York
  - Duke University Medical Center /ID# 234315, Durham, North Carolina
  - Cleveland Clinic Main Campus /ID# 237564, Cleveland, Ohio
- Hospital de Ninos Dr. Orlando Alassia /ID# 235562, Santa Fe, Argentina
- Belarus (3):
  - Grodno Regional Infectious Disease Hospital /ID# 235661, Grodno
  - Mogilev Regional Children's Hospital /ID# 235657, Mogilev
  - Vitebsk Regional Clinical Center for Children /ID# 235659, Vitebsk
- Brazil (2):
  - Duplicate_Hospital Pequeno Princípe /ID# 235629, Curitiba, Paraná
  - Duplicate_Irmandade Santa Casa de Misericórdia de Porto Alegre /ID# 235627, Porto Alegre, Rio Grande do Sul
- Bulgaria (11):
  - University Multiprofile Hospital for Active Treatment Deva Maria EOOD Burgas /ID# 235965, Bulgas
  - MHAT (Multiprofile Hospital for Active Treatment) /ID# 235539, Kozloduy
  - UMHAT Dr Georgi Stranski EAD /ID# 237829, Pleven
  - UMHAT Dr Georgi Stranski EAD /ID# 237830, Pleven
  - Multiprofile Hospital for Active Treatment ( UMHAT) Sveti Georgi EAD Plovdiv /ID# 235487, Plovdiv
  - UMHAT Sveti Georgi /ID# 237026, Plovdiv
  - UMHAT Kanev /ID# 237809, Rousse
  - Medical center 1 Sevlievo /ID# 237470, Sevlievo
  - MHATEM N.I.Pirogov Septic Surgery Clinic /ID# 235541, Sofia
  - SHAT Hematologic Diseases /ID# 237915, Sofia
  - University Multiprofile Hospital for Active Treatment Prof. Dr. Stoyan Kirkovich /ID# 235543, Stara Zagora
- Chile (2):
  - Hospital de Ninos Dr. Roberto del Rio /ID# 235568, Independencia
  - Hospital El Carmen de Maipú /ID# 235570, Santiago
- Colombia (3):
  - Fundacion Cardioinfantil /Id# 238041, Bogota, Cundinamarca
  - Unidad De Investigacion Clinica Universidad De La Sabana /ID# 235566, Chía, Cundinamarca
  - Hospital Universitario San Vic /ID# 238117, Medellín
- Georgia (4):
  - LTD Unimedi Kakheti Batumi Maternal and Child Healthcare Center /ID# 235643, Batumi
  - LEPL Tbilisi State Medical University Givi Zhvania Academic Clinic of Pediatry /ID# 235645, Tbilisi
  - LTD M. Iashvili Children's Central Hospital /ID# 235639, Tbilisi
  - LTD Unimedi Kakheti Children New Hospital /ID# 235634, Tbilisi
- Greece (4):
  - University General Hospital Attikon /ID# 237398, Athens, Attica
  - Papageorgiou General Hospital Thessaloniki /ID# 237505, Stavroupoli (Thessalonikis), Thessaloniki
  - Childrens Hospital of Penteli /ID# 235667, Athens
  - General Hospital of Thessaloniki Hippokrateio /ID# 237186, Thessaloniki
- Guatemala (3):
  - Hospital Valle del Sol /ID# 235569, Guatemala City
  - Hospital Roosevelt /ID# 235520, Guatemala City
  - Hospital del Centro Medico Infectology Department /ID# 235522, Guatemala City
- Latvia (3):
  - Daugavpils Regional Hospital /ID# 237022, Daugavpils
  - Liepaja Regional Hospital /ID# 235650, Liepāja
  - University Childrens Hospital /ID# 235648, Riga
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 236947, Kaunas
  - Klaipeda Children's Hospital /ID# 235652, Klaipėda
  - Duplicate_Children's Hospital Affiliate - Vilnius University Hospital Santariski /ID# 235654, Vilnius
- Mexico (4):
  - Instituto Nacional de Pediatria /ID# 235506, Coyoacán, Mexico City
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez /ID# 237597, Monterrey, Nuevo León
  - Hospital General Dr. Agustin O'Horan /ID# 235510, Mérida, Yucatán
  - Hospital Infantil de Mexico Federico Gomez /ID# 235508, Mexico City
- Panama (2):
  - Hospital Materno Infantil José Domingo de Obaldía /ID# 235625, Chiriquí, Chiriquí Province
  - Hospital Del Niño Dr. José Renán Esquivel /ID# 235572, Panama City
- Poland (3):
  - Wojewodzki Szpital Obserwacyjno-Zakazny im. Tadeusza Browicza /ID# 236920, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Panstwowy Instytut Medyczny MSWiA w Warszawie /ID# 237112, Warsaw, Masovian Voivodeship
  - Specjalistyczny ZOZ nad Matka i Dzieckiem w Poznaniu Oddzial Obserwacyjno /ID# 235518, Poznan
- Romania (4):
  - Institutul National de Boli Infectioase Prof. Dr. Matei Bals /ID# 235606, Sector 2, București
  - Spitalul Clinic de Urgenta pentru Copii ?Louis Turcanu? /ID# 235608, Timișoara, Timiș County
  - Spitalul Clinic de Boli infectioase si Tropicale Dr. Victor Babes /ID# 235610, Bucharest
  - Spitalul Clinic Judeatean Mures /ID# 234728, Târgu Mureş
- Russia (3):
  - Smolensk State Medical University /ID# 236996, Smolensk
  - Stavropol State Medical University /ID# 236239, Stavropol
  - Regional Childrens Hospital /ID# 235560, Vologda
- South Africa (2):
  - Peermed Clinical Trial Centre /ID# 235514, Kempton Park, Gauteng
  - Mzansi Ethical Research Center /ID# 236480, Middelburg, Mpumalanga
- Spain (6):
  - Complejo Hospitalario Universitario de Santiago /ID# 235512, Santiago de Compostela, A Coruna
  - Hospital Sant Joan de Deu /ID# 236797, Esplugues de Llobregat, Barcelona
  - Hospital Donostia /ID# 237773, Donostia / San Sebastian, Guipuzcoa
  - Hospital General Universitario Gregorio Maranon /ID# 236955, Madrid
  - Hospital Universitario La Paz /ID# 237775, Madrid
  - Hospital Universitario y Politecnico La Fe /ID# 237086, Valencia
- Ukraine (6):
  - Ivano-Frankivsk Pediatric Regional Clinical Hospital /ID# 235556, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Dnipropetrovsk Regional children's Clinical Hospital /ID# 235558, Dnipro
  - PE PMC Acinus, Medical and Diagnostic Center /ID# 237514, Kropyvnytskyi
  - Lviv Regional Clinical Hospital /ID# 236921, Lviv
  - Ukrainian Medical Stomatological Academy - Children's City Clinical Hospital /ID# 234886, Poltava
  - Communal Nonprofit Enterprise "Central City Clinical Hospital" of Uzhhorod City /ID# 238058, Uzhhorod

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related info — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intent-to-Treat (ITT) population: all randomized participants
Period: Overall Study
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Started | 91 | 78 | 30
Completed | 91 | 74 | 30
Not Completed | 0 | 4 | 0
Not completed — Withdrawal of consent | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Other, not specified | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: all participants in the ITT population who received at least 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator | Total
Number analyzed (Participants) | 91 | 78 | 30 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.591 (5.4767) | 8.898 (4.9271) | 6.775 (4.2048) | 7.980 (5.1270)
Age, Customized [Count of Participants; unit: Participants]
  Birth to < 3 months (Cohort 5) | 10 | 0 | 0 | 10
  3 months to < 2 years old (Cohort 4) | 9 | 8 | 3 | 20
  2 years to < 6 years old (Cohort 3) | 18 | 17 | 10 | 45
  6 years to < 12 years old (Cohort 2) | 25 | 24 | 11 | 60
  12 years to 17 years old (Cohort 1) | 29 | 29 | 6 | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 25 | 12 | 75
  Male | 53 | 53 | 18 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 1 | 14
  Not Hispanic or Latino | 85 | 71 | 29 | 185
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 1 | 1 | 7
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 6 | 0 | 10
  White | 78 | 69 | 29 | 176
  More than one race | 3 | 1 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Shift From Baseline in Distortion Product Otoacoustic Emission at TOC Visit
Description: Audiologic testing was to be conducted in at least 20 children < 12 years old, of which at least 9 children were < 2 years old. Audiologic testing conducted on infants (< 12 months old) included: evoked otoacoustic emissions testing, acoustic immittance measures (tympanometry and contra and ipsilateral acoustic reflex thresholds) and (optional) threshold auditory brainstem responses. For the older children, testing included evoked otoacoustic emissions testing, acoustic immittance measures (tympanometry and contra ipsilateral acoustic reflex thresholds), and age appropriate behavioral audiologic threshold assessment. Participants with an abnormal audiologic assessment at Day 28 (± 2 days) that exceeded, by a clinically significant margin, any abnormality observed in the Baseline assessment, were considered to have an abnormal audiologic assessment.
Time Frame: Baseline, Day 28 (± 2 days)
Population: Participants who received at least 1 dose of study drug and had baseline and postbaseline values
Measure: Count of Participants; unit: Participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 2 | 0 | 1
Participants
  Baseline & TOC normal | 2 |  | 1
  Baseline normal & TOC abnormal | 0 |  | 0
  Baseline abnormal & TOC normal | 0 |  | 0
  Baseline & TOC abnormal | 0 |  | 0

2. Primary Outcome: Shift From Baseline in Auditory Brainstem Response Test at TOC Visit
Description: as for outcome 1
Time Frame: Baseline, Day 28 (± 2 days)
Population: Participants who received at least 1 dose of study drug and had baseline and postbaseline values
Measure: Count of Participants; unit: Participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 1 | 0 | 0
Participants
  Baseline & TOC normal | 1 |  |
  Baseline normal & TOC abnormal | 0 |  |
  Baseline abnormal & TOC normal | 0 |  |
  Baseline & TOC abnormal | 0 |  |

3. Primary Outcome: Shift From Baseline in Acoustic Immittance Test at TOC Visit
Description: as for outcome 1
Time Frame: Baseline, Day 28 (± 2 days)
Population: Participants who received at least 1 dose of study drug and had baseline and postbaseline values
Measure: Count of Participants; unit: Participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 8 | 4 | 3
Participants
  Baseline & TOC normal | 8 | 4 | 3
  Baseline normal & TOC abnormal | 0 | 0 | 0
  Baseline abnormal & TOC normal | 0 | 0 | 0
  Baseline & TOC abnormal | 0 | 0 | 0

4. Primary Outcome: Shift From Baseline in Behavioral Audiometric Valuation at TOC Visit
Description: as for outcome 1
Time Frame: Baseline, Day 28 (± 2 days)
Population: Participants who received at least 1 dose of study drug and had baseline and postbaseline values
Measure: Count of Participants; unit: Participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 8 | 5 | 4
Participants
  Baseline & TOC normal | 8 | 5 | 4
  Baseline normal & TOC abnormal | 0 | 0 | 0
  Baseline abnormal & TOC normal | 0 | 0 | 0
  Baseline & TOC abnormal | 0 | 0 | 0

5. Primary Outcome: Shift From Baseline in Clostridium Difficile (CD) and Vancomycin-resistant Enterococci (VRE) at TOC Visit
Description: Bowel flora was evaluated in participants from birth to < 2 years of age by performing polymerase chain reaction (PCR) analysis for Clostridium difficile (C diff) and culture for vancomycin-resistant enterococci (VRE) on a stool specimen or rectal swab. Samples were analyzed at Baseline and at the Test of Cure (TOC) visit.
Time Frame: Baseline, Day 28 (± 2 days)
Population: Participants aged birth to < 2 years who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Groups:
- Dalbavancin Single-dose: Participants received dalbavancin administered intravenously as follows: birth to < 3 months of age and 3 months to < 6 years old: 22.5 mg/kg (maximum 1500 mg) on Day 1; ≥6 years to 17 years old (inclusive): 18 mg/kg (maximum 1500 mg) on Day 1.
- Comparator: Participants 3 months to < 6 years old and ≥6 years to 17 years old (inclusive) who were randomized to the comparator arm received a 10-14 day course of either vancomycin 10 to 15 mg/kg/dose, not to exceed a total daily dose of 4000 mg; or oxacillin 30 mg/kg/dose or flucloxacillin 50 mg/kg/dose, not to exceed a total daily dose of 2000 mg. Based on local practice patterns and approvals for clinical use in the pediatric population, oxacillin or flucloxacillin were supplied as an IV comparator.
  Those on oxacillin or flucloxacillin were permitted to switch to oral cefadroxil (dose for infants and children: 15 mg/kg/dose every 12 hours, maximum 2 g/day; dose for adolescents: 500-1000 mg every 12 hours), and if infection with methicillin-resistant S. aureus was documented, they were allowed to switch from IV vancomycin to oral therapy with clindamycin 10 mg/kg every 8 hours at the discretion of the investigator after at least 72 hours of IV therapy.
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 19 | 8 | 3
Participants
  C diff Baseline & TOC positive | 1 | 0 | 0
  C diff Baseline positive & TOC negative | 3 | 1 | 0
  C diff Baseline positive & TOC missing | 2 | 1 | 0
  C diff Baseline negative & TOC positive | 0 | 0 | 0
  C diff Baseline negative & TOC negative | 10 | 4 | 1
  C diff Baseline negative & TOC missing | 1 | 1 | 0
  C diff Baseline missing & TOC positive | 0 | 0 | 0
  C diff Baseline missing & TOC negative | 2 | 0 | 1
  C diff Baseline missing & TOC missing | 0 | 1 | 1
  VRE Baseline & TOC positive | 1 | 0 | 0
  VRE Baseline positive & TOC negative | 0 | 0 | 0
  VRE Baseline positive & TOC missing | 0 | 1 | 0
  VRE Baseline negative & TOC positive | 0 | 0 | 0
  VRE Baseline negative & TOC negative | 15 | 5 | 0
  VRE Baseline negative & TOC missing | 1 | 2 | 2
  VRE Baseline missing & TOC positive | 1 | 0 | 0
  VRE Baseline missing & TOC negative | 1 | 0 | 1
  VRE Baseline missing & TOC missing | 0 | 0 | 0

6. Secondary Outcome: Clinical Response at 48-72 Hours
Description: Clinical response defined as ≥20% reduction in lesion size compared to Baseline in Cohorts 1-4; cessation of increase in lesion size and decreased erythema or tenderness compared to Baseline with no appearance of new lesions in those with ABSSSI in Cohort 5; and improvement of at least one abnormal clinical and laboratory parameter related to sepsis in those diagnosed with sepsis in Cohort 5. To be considered a clinical responder, participants must have been alive and not have received rescue therapy.
  Presented for the modified intent-to-treat (mITT) population: all participants who received at least one dose of study drug and had a diagnosis of ABSSSI (or a suspected or confirmed sepsis for those in Cohort 5) not known to be caused exclusively by a Gram-negative organism.
Time Frame: Baseline, 48-72 hours
Population: Participants in the mITT population with non-missing analysis values at the visit
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 85 | 74 | 29
percentage of participants
  Clinical Responder | 96.5 | 98.6 | 89.7
  Clinical Non-Responder | 3.5 | 1.4 | 10.3

7. Secondary Outcome: Clinical Response at the End of Treatment (EOT) Visit (Investigator Assessment of Clinical Outcome)
Description: Cure: Resolution of clinical signs and symptoms of infection (CSSI) compared to Baseline. No additional antibacterial Tx required for disease under study.
  Improvement: For Cohorts 1-4 and Cohort 5 with ABSSSI, reduction in severity of ≥2, but not all CSSI, when compared with Baseline. For Cohort 5 with sepsis, reduction in severity of ≥1 abnormal clinical and laboratory parameter related to sepsis, when compared with Baseline. For Cohorts 1-4, no additional antibacterial Tx required for disease under study. For Cohort 5, no rescue antibiotics required after ≥48 hours of start of study Tx.
  Failure: Persistence or progression of Baseline CSSI after 48 hours of Tx OR development of new findings consistent with active infection.
  Unknown: Extenuating circumstances precluding classification to Cure, Improvement, or Failure.
  Presented for the modified intent-to-treat (mITT) population.
Time Frame: Baseline, Day 14 (± 2 Days)
Population: Participants in the mITT population with non-missing analysis values at the visit
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 84 | 73 | 29
percentage of participants
  Clinical Cure | 92.9 | 93.2 | 100
  Improvement | 6.0 | 5.5 | 0
  Clinical Failure | 1.2 | 1.4 | 0
  Unknown | 0 | 0 | 0

8. Secondary Outcome: Clinical Response at the End of Treatment (EOT) Visit (Clinical Response by Sponsor)
Description: Definitions used for the Sponsor assessment were the same as those used for the Investigator assessment. The occurrence of any of the following conditions resulted in reassignment by the Sponsor to clinical failure: 1) assessment of clinical failure at a previous time point, 2) Cohorts 1-4: receipt of concomitant antibiotic with activity against participant's isolate of disease under study prior to evaluation time point; Cohort 5: receipt of rescue therapy (additional antibiotic therapy initiated ≥48 hrs after study drug start), 3) unplanned surgical procedure (e.g., incision and drainage of abscess, major debridement, amputation) for non-improving or worsening infection after 72 hrs of study drug treatment.
  Presented for the modified intent-to-treat (mITT) population: all participants who received ≥1 dose of study drug and had a diagnosis of ABSSSI (or a suspected or confirmed sepsis for those in Cohort 5) not known to be caused exclusively by a Gram-negative organism.
Time Frame: Baseline, Day 14 (± 2 Days)
Population: Participants in the mITT population with non-missing analysis values at the visit
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 84 | 74 | 30
percentage of participants
  Cure | 90.5 | 91.9 | 100
  Improvement | 7.1 | 5.4 | 0
  Failure | 2.4 | 2.7 | 0
  Unknown | 0 | 0 | 0

9. Secondary Outcome: Clinical Response at the Test of Cure (TOC) Visit (Investigator Assessment of Clinical Outcome)
Description: Cure: Resolution of clinical signs and symptoms of infection (CSSI) compared to Baseline. No additional antibacterial Tx required for disease under study.
  Failure: Persistence or progression of Baseline CSSI after 48 hours of Tx OR development of new findings consistent with active infection.
  Unknown: Extenuating circumstances precluding classification to Cure or Failure.
  Presented for the modified intent-to-treat (mITT) population.
Time Frame: Baseline, Day 28 (± 2 Days)
Population: Participants in the mITT population with non-missing analysis values at the visit
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 83 | 73 | 30
percentage of participants
  Clinical Cure | 98.8 | 98.6 | 100
  Clinical Failure | 1.2 | 1.4 | 0
  Unknown | 0 | 0 | 0

10. Secondary Outcome: Clinical Response at the Test of Cure (TOC) Visit (Clinical Response by Sponsor)
Description: as for outcome 8
Time Frame: Baseline, Day 28 (± 2 Days)
Population: Participants in the mITT population with non-missing analysis values at the visit
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 83 | 74 | 30
percentage of participants
  Cure | 95.2 | 97.3 | 100
  Failure | 2.4 | 2.7 | 0
  Unknown | 2.4 | 0 | 0

11. Secondary Outcome: Clinical Response at the Follow-Up Visit (Investigator Assessment of Clinical Outcome)
Description: as for outcome 9
Time Frame: Baseline, Day 54 (± 7 days)
Population: Participants in the mITT population with non-missing analysis values at the visit
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 85 | 73 | 30
percentage of participants
  Clinical Cure | 97.6 | 97.3 | 100
  Clinical Failure | 1.2 | 1.4 | 0
  Unknown | 1.2 | 1.4 | 0

12. Secondary Outcome: Clinical Response at the Follow-Up Visit (Clinical Response by Sponsor)
Description: as for outcome 8
Time Frame: Baseline, Day 54 (± 7 days)
Population: Participants in the mITT population with non-missing analysis values at the visit
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 84 | 73 | 30
percentage of participants
  Cure | 96.4 | 97.3 | 100
  Failure | 2.4 | 2.7 | 0
  Unknown | 1.2 | 0 | 0

13. Secondary Outcome: Clinical Response by Baseline Pathogen at 48-72 Hours (Clinical Response by Sponsor)
Description: Clinical response defined as ≥20% reduction in lesion size compared to Baseline in Cohorts 1-4; cessation of increase in lesion size and decreased erythema or tenderness compared to Baseline with no appearance of new lesions in those with ABSSSI in Cohort 5; and improvement of at least one abnormal clinical and laboratory parameter related to sepsis in those diagnosed with sepsis in Cohort 5. To be considered a clinical responder, participants must have been alive and not have received rescue therapy.
  Presented for the microbiological intent-to-treat (microITT) population: all randomized (or enrolled in Cohort 5) participants who had at least 1 Gram-positive pathogen isolated at Baseline.
Time Frame: Baseline, 48-72 hours
Population: Participants in the microITT population with specified baseline pathogen
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 52 | 55 | 18
percentage of participants
  S. aureus (MRSA),Clinical Responder: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Clinical Responder | 100 | 100 |
  S. aureus (MRSA),Clinical Non-Responder: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Clinical Non-Responder | 0 | 0 |
  S. aureus (MSSA),Clinical Responder: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Clinical Responder | 97.9 | 95.5 | 85.7
  S. aureus (MSSA),Clinical Non-Responder: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Clinical Non-Responder | 2.1 | 2.3 | 7.1
  S. aureus (MSSA),Missing: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Missing | 0 | 2.3 | 7.1
  S. agalactiae, Clinical Responder: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Clinical Responder |  | 100 |
  S. agalactiae, Clinical Non-Responder: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Clinical Non-Responder |  | 0 |
  S. anginosus, Clinical Responder: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Clinical Responder | 100 |  |
  S. anginosus, Clinical Non-Responder: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Clinical Non-Responder | 0 |  |
  S. constellatus, Clinical Responder: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Clinical Responder |  | 100 |
  S. constellatus, Clinical Non-Responder: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Clinical Non-Responder |  | 0 |
  S. intermedius, Clinical Responder: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Clinical Responder |  | 100 |
  S. intermedius, Clinical Non-Responder: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Clinical Non-Responder |  | 0 |
  S. pyogenes, Clinical Responder: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Clinical Responder | 80 | 75 | 100
  S. pyogenes, Clinical Non-Responder: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Clinical Non-Responder | 20 | 0 | 0
  S. pyogenes, Missing: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Missing | 0 | 25 | 0
  E. faecalis, Clinical Responder: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Clinical Responder | 100 | 100 |
  E. faecalis, Clinical Non-Responder: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Clinical Non-Responder | 0 | 0 |

14. Secondary Outcome: Clinical Response by Baseline Pathogen at the End of Treatment (EOT) Visit (Investigator Assessment of Clinical Outcome)
Description: Cure: Resolution of clinical signs/symptoms of infection (CSSI) compared to Baseline. No additional antibacterial Tx required for disease under study.
  Improvement: Cohorts 1-4 and Cohort 5 with ABSSSI: reduction in severity of ≥2, but not all CSSI, when compared to Baseline. Cohort 5 with sepsis: reduction in severity of ≥1 abnormal clinical/laboratory parameter related to sepsis, when compared to Baseline. Cohorts 1-4: no additional antibacterial Tx required for disease under study. Cohort 5: no rescue antibiotics required after ≥48 hrs of start of study Tx.
  Failure: Persistence/progression of Baseline CSSI after 48 hrs of Tx OR development of new findings consistent with active infection.
  Unknown: Extenuating circumstances precluding classification to Cure, Improvement, or Failure.
  Presented for the microbiological intent-to-treat (microITT) population: all randomized (or enrolled in Cohort 5) participants who had at least 1 Gram-positive pathogen isolated at Baseline.
Time Frame: Baseline, Day 14 (± 2 Days)
Population: Participants in the microITT population with specified baseline pathogen
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 52 | 55 | 18
percentage of participants
  S. aureus (MRSA),Clinical Cure: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Clinical Cure | 100 | 75 |
  S. aureus (MRSA),Improvement: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Improvement | 0 | 0 |
  S. aureus (MRSA),Clinical Failure: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Clinical Failure | 0 | 0 |
  S. aureus (MRSA),Unknown: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Unknown | 0 | 0 |
  S. aureus (MRSA),Missing: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Missing | 0 | 25 |
  S. aureus (MSSA),Clinical Cure: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Clinical Cure | 91.5 | 86.4 | 100
  S. aureus (MSSA),Improvement: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Improvement | 4.3 | 4.5 | 0
  S. aureus (MSSA),Clinical Failure: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Clinical Failure | 2.1 | 2.3 | 0
  S. aureus (MSSA),Unknown: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Unknown | 0 | 0 | 0
  S. aureus (MSSA),Missing: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Missing | 2.1 | 6.8 | 0
  S. agalactiae, Clinical Cure: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Clinical Cure |  | 100 |
  S. agalactiae, Improvement: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Improvement |  | 0 |
  S. agalactiae, Clinical Failure: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Clinical Failure |  | 0 |
  S. agalactiae, Unknown: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Unknown |  | 0 |
  S. anginosus, Clinical Cure: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Clinical Cure | 100 |  |
  S. anginosus, Improvement: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Improvement | 0 |  |
  S. anginosus, Clinical Failure: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Clinical Failure | 0 |  |
  S. anginosus, Unknown: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Unknown | 0 |  |
  S. constellatus, Clinical Cure: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Clinical Cure |  | 100 |
  S. constellatus, Improvement: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Improvement |  | 0 |
  S. constellatus, Clinical Failure: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Clinical Failure |  | 0 |
  S. constellatus, Unknown: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Unknown |  | 0 |
  S. intermedius, Clinical Cure: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Clinical Cure |  | 100 |
  S. intermedius, Improvement: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Improvement |  | 0 |
  S. intermedius, Clinical Failure: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Clinical Failure |  | 0 |
  S. intermedius, Unknown: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Unknown |  | 0 |
  S. pyogenes, Clinical Cure: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Clinical Cure | 80 | 50 | 100
  S. pyogenes, Improvement: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Improvement | 0 | 25 | 0
  S. pyogenes, Clinical Failure: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Clinical Failure | 20 | 0 | 0
  S. pyogenes, Unknown: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Unknown | 0 | 0 | 0
  S. pyogenes, Missing: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Missing | 0 | 25 | 0
  E. faecalis, Clinical Cure: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Clinical Cure | 100 | 100 |
  E. faecalis, Improvement: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Improvement | 0 | 0 |
  E. faecalis, Clinical Failure: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Clinical Failure | 0 | 0 |
  E. faecalis, Unknown: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Unknown | 0 | 0 |

15. Secondary Outcome: Clinical Response by Baseline Pathogen at the End of Treatment (EOT) Visit (Clinical Response by Sponsor)
Description: Definitions used for the Sponsor assessment were the same as those used for the Investigator assessment. The occurrence of any of the following conditions resulted in reassignment by the Sponsor to clinical failure: 1) assessment of clinical failure at a previous time point, 2) Cohorts 1-4: receipt of concomitant antibiotic with activity against participant's isolate of disease under study prior to evaluation time point; Cohort 5: receipt of rescue therapy (additional antibiotic therapy initiated ≥48 hrs after study drug start), 3) unplanned surgical procedure (e.g., incision and drainage of abscess, major debridement, amputation) for non-improving or worsening infection after 72 hrs of study drug treatment.
  Presented for the microbiological intent-to-treat (microITT) population: all randomized (or enrolled in Cohort 5) participants who had at least 1 Gram-positive pathogen isolated at Baseline.
Time Frame: Baseline, Day 14 (± 2 Days)
Population: Participants in the microITT population with specified baseline pathogen
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 52 | 55 | 18
percentage of participants
  S. aureus (MRSA),Cure: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Cure | 100 | 75 |
  S. aureus (MRSA),Improvement: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Improvement | 0 | 0 |
  S. aureus (MRSA),Failure: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Failure | 0 | 25 |
  S. aureus (MRSA),Unknown: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Unknown | 0 | 0 |
  S. aureus (MSSA),Cure: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Cure | 91.5 | 86.4 | 100
  S. aureus (MSSA),Improvement: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Improvement | 4.3 | 4.5 | 0
  S. aureus (MSSA),Failure: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Failure | 2.1 | 4.5 | 0
  S. aureus (MSSA),Unknown: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Unknown | 0 | 0 | 0
  S. aureus (MSSA),Missing: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Missing | 2.1 | 4.5 | 0
  S. agalactiae, Cure: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Cure |  | 100 |
  S. agalactiae, Improvement: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Improvement |  | 0 |
  S. agalactiae, Failure: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Failure |  | 0 |
  S. agalactiae, Unknown: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Unknown |  | 0 |
  S. anginosus, Cure: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Cure | 100 |  |
  S. anginosus, Improvement: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Improvement | 0 |  |
  S. anginosus, Failure: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Failure | 0 |  |
  S. anginosus, Unknown: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Unknown | 0 |  |
  S. constellatus, Cure: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Cure |  | 100 |
  S. constellatus, Improvement: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Improvement |  | 0 |
  S. constellatus, Failure: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Failure |  | 0 |
  S. constellatus, Unknown: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Unknown |  | 0 |
  S. intermedius, Cure: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Cure |  | 100 |
  S. intermedius, Improvement: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Improvement |  | 0 |
  S. intermedius, Failure: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Failure |  | 0 |
  S. intermedius, Unknown: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Unknown |  | 0 |
  S. pyogenes, Cure: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Cure | 80 | 50 | 100
  S. pyogenes, Improvement: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Improvement | 0 | 25 | 0
  S. pyogenes, Failure: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Failure | 20 | 0 | 0
  S. pyogenes, Unknown: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Unknown | 0 | 0 | 0
  S. pyogenes, Missing: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Missing | 0 | 25 | 0
  E. faecalis, Cure: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Cure | 100 | 100 |
  E. faecalis, Improvement: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Improvement | 0 | 0 |
  E. faecalis, Failure: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Failure | 0 | 0 |
  E. faecalis, Unknown: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Unknown | 0 | 0 |

16. Secondary Outcome: Clinical Response by Baseline Pathogen at the Test of Cure (TOC) Visit (Investigator Assessment of Clinical Outcome)
Description: Cure: Resolution of clinical signs and symptoms of infection (CSSI) compared to Baseline. No additional antibacterial Tx required for disease under study.
  Failure: Persistence or progression of Baseline CSSI after 48 hours of Tx OR development of new findings consistent with active infection.
  Unknown: Extenuating circumstances precluding classification to Cure or Failure.
  Presented for the microbiological intent-to-treat (microITT) population: all randomized (or enrolled in Cohort 5) participants who had at least 1 Gram-positive pathogen isolated at Baseline.
Time Frame: Baseline, Day 28 (± 2 Days)
Population: Participants in the microITT population with specified baseline pathogen
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 52 | 55 | 18
percentage of participants
  S. aureus (MRSA),Clinical Cure: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Clinical Cure | 100 | 75 |
  S. aureus (MRSA),Clinical Failure: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Clinical Failure | 0 | 0 |
  S. aureus (MRSA),Unknown: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Unknown | 0 | 0 |
  S. aureus (MRSA),Missing: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Missing | 0 | 25 |
  S. aureus (MSSA),Clinical Cure: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Clinical Cure | 95.7 | 90.9 | 100
  S. aureus (MSSA),Clinical Failure: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Clinical Failure | 2.1 | 2.3 | 0
  S. aureus (MSSA),Unknown: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Unknown | 0 | 0 | 0
  S. aureus (MSSA),Missing: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Missing | 2.2 | 6.8 | 0
  S. agalactiae, Clinical Cure: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Clinical Cure |  | 100 |
  S. agalactiae, Clinical Failure: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Clinical Failure |  | 0 |
  S. agalactiae, Unknown: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Unknown |  | 0 |
  S. anginosus, Clinical Cure: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Clinical Cure | 100 |  |
  S. anginosus, Clinical Failure: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Clinical Failure | 0 |  |
  S. anginosus, Unknown: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Unknown | 0 |  |
  S. constellatus, Clinical Cure: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Clinical Cure |  | 100 |
  S. constellatus, Clinical Failure: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Clinical Failure |  | 0 |
  S. constellatus, Unknown: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Unknown |  | 0 |
  S. intermedius, Clinical Cure: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Clinical Cure |  | 100 |
  S. intermedius, Clinical Failure: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Clinical Failure |  | 0 |
  S. intermedius, Unknown: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Unknown |  | 0 |
  S. pyogenes, Clinical Cure: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Clinical Cure | 80 | 75 | 100
  S. pyogenes, Clinical Failure: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Clinical Failure | 20 | 0 | 0
  S. pyogenes, Unknown: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Unknown | 0 | 0 | 0
  S. pyogenes, Missing: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Missing | 0 | 25 | 0
  E. faecalis, Clinical Cure: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Clinical Cure | 100 | 100 |
  E. faecalis, Clinical Failure: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Clinical Failure | 0 | 0 |
  E. faecalis, Unknown: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Unknown | 0 | 0 |

17. Secondary Outcome: Clinical Response by Baseline Pathogen at the Test of Cure (TOC) Visit (Clinical Response by Sponsor)
Description: as for outcome 15
Time Frame: Baseline, Day 28 (± 2 Days)
Population: Participants in the microITT population with specified baseline pathogen
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 52 | 55 | 18
percentage of participants
  S. aureus (MRSA),Cure: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Cure | 100 | 75 |
  S. aureus (MRSA),Failure: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Failure | 0 | 25 |
  S. aureus (MRSA),Unknown: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Unknown | 0 | 0 |
  S. aureus (MSSA),Cure: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Cure | 91.5 | 90.9 | 100
  S. aureus (MSSA),Failure: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Failure | 2.1 | 4.5 | 0
  S. aureus (MSSA),Unknown: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Unknown | 4.3 | 0 | 0
  S. aureus (MSSA),Missing: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Missing | 2.1 | 4.5 | 0
  S. agalactiae, Cure: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Cure |  | 100 |
  S. agalactiae, Failure: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Failure |  | 0 |
  S. agalactiae, Unknown: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Unknown |  | 0 |
  S. anginosus, Cure: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Cure | 100 |  |
  S. anginosus, Failure: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Failure | 0 |  |
  S. anginosus, Unknown: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Unknown | 0 |  |
  S. constellatus, Cure: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Cure |  | 100 |
  S. constellatus, Failure: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Failure |  | 0 |
  S. constellatus, Unknown: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Unknown |  | 0 |
  S. intermedius, Cure: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Cure |  | 100 |
  S. intermedius, Failure: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Failure |  | 0 |
  S. intermedius, Unknown: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Unknown |  | 0 |
  S. pyogenes, Cure: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Cure | 80 | 75 | 100
  S. pyogenes, Failure: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Failure | 20 | 0 | 0
  S. pyogenes, Unknown: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Unknown | 0 | 0 | 0
  S. pyogenes, Missing: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Missing | 0 | 25 | 0
  E. faecalis, Cure: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Cure | 100 | 100 |
  E. faecalis, Failure: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Failure | 0 | 0 |
  E. faecalis, Unknown: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Unknown | 0 | 0 |

18. Secondary Outcome: Clinical Response by Baseline Pathogen at the Follow-up Visit (Investigator Assessment of Clinical Outcome)
Description: as for outcome 16
Time Frame: Baseline, Day 54 (± 7 days)
Population: Participants in the microITT population with specified baseline pathogen
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 52 | 55 | 18
percentage of participants
  S. aureus (MRSA),Clinical Cure: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Clinical Cure | 50 | 50 |
  S. aureus (MRSA),Clinical Failure: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Clinical Failure | 0 | 0 |
  S. aureus (MRSA),Unknown: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Unknown | 50 | 25 |
  S. aureus (MRSA),Missing: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Missing | 0 | 25 |
  S. aureus (MSSA),Clinical Cure: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Clinical Cure | 95.7 | 88.6 | 100
  S. aureus (MSSA),Clinical Failure: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Clinical Failure | 2.1 | 2.3 | 0
  S. aureus (MSSA),Unknown: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Unknown | 2.1 | 0 | 0
  S. aureus (MSSA),Missing: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Missing | 0 | 9.1 | 0
  S. agalactiae, Clinical Cure: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Clinical Cure |  | 100 |
  S. agalactiae, Clinical Failure: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Clinical Failure |  | 0 |
  S. agalactiae, Unknown: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Unknown |  | 0 |
  S. anginosus, Clinical Cure: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Clinical Cure | 100 |  |
  S. anginosus, Clinical Failure: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Clinical Failure | 0 |  |
  S. anginosus, Unknown: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Unknown | 0 |  |
  S. constellatus, Clinical Cure: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Clinical Cure |  | 100 |
  S. constellatus, Clinical Failure: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Clinical Failure |  | 0 |
  S. constellatus, Unknown: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Unknown |  | 0 |
  S. intermedius, Clinical Cure: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Clinical Cure |  | 100 |
  S. intermedius, Clinical Failure: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Clinical Failure |  | 0 |
  S. intermedius, Unknown: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Unknown |  | 0 |
  S. pyogenes, Clinical Cure: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Clinical Cure | 80 | 75 | 100
  S. pyogenes, Clinical Failure: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Clinical Failure | 20 | 0 | 0
  S. pyogenes, Unknown: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Unknown | 0 | 0 | 0
  S. pyogenes, Missing: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Missing | 0 | 25 | 0
  E. faecalis, Clinical Cure: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Clinical Cure | 100 | 100 |
  E. faecalis, Clinical Failure: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Clinical Failure | 0 | 0 |
  E. faecalis, Unknown: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Unknown | 0 | 0 |

19. Secondary Outcome: Clinical Response by Baseline Pathogen at the Follow-up Visit (Clinical Response by Sponsor)
Description: as for outcome 15
Time Frame: Baseline, Day 54 (± 7 days)
Population: Participants in the microITT population with specified baseline pathogen
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 52 | 55 | 18
percentage of participants
  S. aureus (MRSA),Cure: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Cure | 50 | 50 |
  S. aureus (MRSA),Failure: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Failure | 0 | 25 |
  S. aureus (MRSA),Unknown: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Unknown | 0 | 0 |
  S. aureus (MRSA),Missing: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA),Missing | 50 | 25 |
  S. aureus (MSSA),Cure: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Cure | 93.6 | 88.6 | 100
  S. aureus (MSSA),Failure: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Failure | 2.1 | 4.5 | 0
  S. aureus (MSSA),Unknown: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Unknown | 2.1 | 0 | 0
  S. aureus (MSSA),Missing: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA),Missing | 2.1 | 6.8 | 0
  S. agalactiae, Cure: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Cure |  | 100 |
  S. agalactiae, Failure: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Failure |  | 0 |
  S. agalactiae, Unknown: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Unknown |  | 0 |
  S. anginosus, Cure: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Cure | 100 |  |
  S. anginosus, Failure: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Failure | 0 |  |
  S. anginosus, Unknown: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Unknown | 0 |  |
  S. constellatus, Cure: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Cure |  | 100 |
  S. constellatus, Failure: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Failure |  | 0 |
  S. constellatus, Unknown: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Unknown |  | 0 |
  S. intermedius, Cure: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Cure |  | 100 |
  S. intermedius, Failure: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Failure |  | 0 |
  S. intermedius, Unknown: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Unknown |  | 0 |
  S. pyogenes, Cure: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Cure | 80 | 75 | 100
  S. pyogenes, Failure: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Failure | 20 | 0 | 0
  S. pyogenes, Unknown: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Unknown | 0 | 0 | 0
  S. pyogenes, Missing: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Missing | 0 | 25 | 0
  E. faecalis, Cure: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Cure | 100 | 100 |
  E. faecalis, Failure: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Failure | 0 | 0 |
  E. faecalis, Unknown: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Unknown | 0 | 0 |

20. Secondary Outcome: Microbiological Response at 48-72 Hours
Description: Eradication: Source specimen demonstrated absence of the original Baseline pathogen.
  Presumed eradication: Source specimen was not available to culture and the participant was assessed as a clinical responder.
  Persistence: Source specimen demonstrated continued presence of the original Baseline pathogen.
  Presumed persistence: Source specimen was not available to culture and the participant was assessed as a clinical non-responder.
  Indeterminate: Source specimen was not available to culture and the participant's clinical response was unknown or missing.
  Presented for the microbiological intent-to-treat (microITT) population: all randomized (or enrolled in Cohort 5) participants who had at least 1 Gram-positive pathogen isolated at Baseline.
Time Frame: Baseline, 48-72 hours
Population: Participants in the microITT population with non-missing analysis values at the visit
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 52 | 54 | 18
percentage of participants
  Eradication | 0 | 1.9 | 0
  Presumed eradication | 98.1 | 94.4 | 88.9
  Persistence | 0 | 1.9 | 0
  Presumed persistence | 1.9 | 1.9 | 5.6
  Indeterminate | 0 | 0 | 5.6

21. Secondary Outcome: Microbiological Response at the End of Treatment (EOT) Visit
Description: Eradication: Source specimen demonstrated absence of the original Baseline pathogen.
  Presumed eradication: Source specimen was not available to culture and the participant was assessed as a clinical cure or improvement.
  Persistence: Source specimen demonstrated continued presence of the original Baseline pathogen.
  Presumed persistence: Source specimen was not available to culture and the participant was assessed as a clinical failure.
  Indeterminate: Source specimen was not available to culture and the participant's clinical response was unknown or missing.
  Presented for the microbiological intent-to-treat (microITT) population: all randomized (or enrolled in Cohort 5) participants who had at least 1 Gram-positive pathogen isolated at Baseline.
Time Frame: Baseline, Day 14 (± 2 Days)
Population: Participants in the microITT population with non-missing analysis values at the visit
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 52 | 54 | 18
percentage of participants
  Eradication | 0 | 1.9 | 0
  Presumed eradication | 96.2 | 92.6 | 100
  Persistence | 0 | 1.9 | 0
  Presumed persistence | 1.9 | 1.9 | 0
  Indeterminate | 1.9 | 1.9 | 0

22. Secondary Outcome: Microbiological Response at the Test of Cure (TOC) Visit
Description: Eradication: Source specimen demonstrated absence of the original Baseline pathogen.
  Presumed eradication: Source specimen was not available to culture and the participant was assessed as a clinical cure.
  Persistence: Source specimen demonstrated continued presence of the original Baseline pathogen.
  Presumed persistence: Source specimen was not available to culture and the participant was assessed as a clinical failure.
  Indeterminate: Source specimen was not available to culture and the participant's clinical response was unknown or missing.
  Presented for the microbiological intent-to-treat (microITT) population: all randomized (or enrolled in Cohort 5) participants who had at least 1 Gram-positive pathogen isolated at Baseline.
Time Frame: Baseline, Day 28 (± 2 Days)
Population: Participants in the microITT population with non-missing analysis values at the visit
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 52 | 54 | 18
percentage of participants
  Eradication | 0 | 1.9 | 0
  Presumed eradication | 92.3 | 92.6 | 100
  Persistence | 0 | 0 | 0
  Presumed persistence | 1.9 | 3.7 | 0
  Indeterminate | 5.8 | 1.9 | 0

23. Secondary Outcome: Microbiological Response at the Follow-Up Visit
Description: as for outcome 22
Time Frame: Baseline, Day 54 (± 7 days)
Population: Participants in the microITT population with non-missing analysis values at the visit
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 52 | 54 | 18
percentage of participants
  Eradication | 0 | 1.9 | 0
  Presumed eradication | 94.2 | 88.9 | 100
  Persistence | 0 | 0 | 0
  Presumed persistence | 1.9 | 3.7 | 0
  Indeterminate | 3.8 | 5.6 | 0

24. Secondary Outcome: Microbiological Response at 48-72 Hours by Baseline Gram-positive Pathogen
Description: Eradication: Source specimen demonstrated absence of the original Baseline pathogen.
  Presumed eradication: Source specimen was not available to culture and the participant was assessed as a clinical responder.
  Persistence: Source specimen demonstrated continued presence of the original Baseline pathogen.
  Presumed persistence: Source specimen was not available to culture and the participant was assessed as a clinical non-responder.
  Indeterminate: Source specimen was not available to culture and the participant's clinical response was unknown or missing.,
  Presented for the microbiological intent-to-treat (microITT) population: all randomized (or enrolled in Cohort 5) participants who had at least 1 Gram-positive pathogen isolated at Baseline.
Time Frame: Baseline, 48-72 hours
Population: Participants in the microITT population with specified baseline pathogen
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 52 | 55 | 18
percentage of participants
  S. aureus (MRSA), Eradication: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA), Eradication | 0 | 0 |
  S. aureus (MRSA), Presumed eradication: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA), Presumed eradication | 100 | 100 |
  S. aureus (MRSA), Persistence: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA), Persistence | 0 | 0 |
  S. aureus (MRSA), Presumed persistence: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA), Presumed persistence | 0 | 0 |
  S. aureus (MRSA), Indeterminate: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA), Indeterminate | 0 | 0 |
  S. aureus (MSSA), Eradication: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Eradication | 0 | 2.3 | 0
  S. aureus (MSSA), Presumed eradication: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Presumed eradication | 97.9 | 90.9 | 85.7
  S. aureus (MSSA), Persistence: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Persistence | 0 | 2.3 | 0
  S. aureus (MSSA), Presumed persistence: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Presumed persistence | 2.1 | 2.3 | 7.1
  S. aureus (MSSA), Indeterminate: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Indeterminate | 0 | 0 | 7.1
  S. aureus (MSSA), Missing: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Missing | 0 | 2.3 | 0
  S. agalactiae, Eradication: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Eradication |  | 0 |
  S. agalactiae, Presumed eradication: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Presumed eradication |  | 100 |
  S. agalactiae, Persistence: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Persistence |  | 0 |
  S. agalactiae, Presumed persistence: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Presumed persistence |  | 0 |
  S. agalactiae, Indeterminate: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Indeterminate |  | 0 |
  S. anginosus, Eradication: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Eradication | 0 |  |
  S. anginosus, Presumed eradication: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Presumed eradication | 100 |  |
  S. anginosus, Persistence: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Persistence | 0 |  |
  S. anginosus, Presumed persistence: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Presumed persistence | 0 |  |
  S. anginosus, Indeterminate: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Indeterminate | 0 |  |
  S. constellatus, Eradication: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Eradication |  | 0 |
  S. constellatus, Presumed eradication: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Presumed eradication |  | 100 |
  S. constellatus, Persistence: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Persistence |  | 0 |
  S. constellatus, Presumed persistence: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Presumed persistence |  | 0 |
  S. constellatus, Indeterminate: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Indeterminate |  | 0 |
  S. intermedius, Eradication: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Eradication |  | 0 |
  S. intermedius, Presumed eradication: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Presumed eradication |  | 100 |
  S. intermedius, Persistence: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Persistence |  | 0 |
  S. intermedius, Presumed persistence: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Presumed persistence |  | 0 |
  S. intermedius, Indeterminate: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Indeterminate |  | 0 |
  S. mitis/oralis, Eradication: number analyzed (Participants) | 1 | 1 | 1
  S. mitis/oralis, Eradication | 0 | 0 | 0
  S. mitis/oralis, Presumed eradication: number analyzed (Participants) | 1 | 1 | 1
  S. mitis/oralis, Presumed eradication | 100 | 100 | 100
  S. mitis/oralis, Persistence: number analyzed (Participants) | 1 | 1 | 1
  S. mitis/oralis, Persistence | 0 | 0 | 0
  S. mitis/oralis, Presumed persistence: number analyzed (Participants) | 1 | 1 | 1
  S. mitis/oralis, Presumed persistence | 0 | 0 | 0
  S. mitis/oralis, Indeterminate: number analyzed (Participants) | 1 | 1 | 1
  S. mitis/oralis, Indeterminate | 0 | 0 | 0
  S. pyogenes, Eradication: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Eradication | 0 | 0 | 0
  S. pyogenes, Presumed eradication: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Presumed eradication | 80 | 75 | 100
  S. pyogenes, Persistence: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Persistence | 0 | 0 | 0
  S. pyogenes, Presumed persistence: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Presumed persistence | 20 | 0 | 0
  S. pyogenes, Indeterminate: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Indeterminate | 0 | 0 | 0
  S. pyogenes, Missing: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Missing | 0 | 25 | 0
  E. faecalis, Eradication: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Eradication | 0 | 0 |
  E. faecalis, Presumed eradication: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Presumed eradication | 100 | 100 |
  E. faecalis, Persistence: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Persistence | 0 | 0 |
  E. faecalis, Presumed persistence: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Presumed persistence | 0 | 0 |
  E. faecalis, Indeterminate: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Indeterminate | 0 | 0 |
  E. hirae, Eradication: number analyzed (Participants) | 1 | 0 | 0
  E. hirae, Eradication | 0 |  |
  E. hirae, Presumed eradication: number analyzed (Participants) | 1 | 0 | 0
  E. hirae, Presumed eradication | 100 |  |
  E. hirae, Persistence: number analyzed (Participants) | 1 | 0 | 0
  E. hirae, Persistence | 0 |  |
  E. hirae, Presumed persistence: number analyzed (Participants) | 1 | 0 | 0
  E. hirae, Presumed persistence | 0 |  |
  E. hirae, Indeterminate: number analyzed (Participants) | 1 | 0 | 0
  E. hirae, Indeterminate | 0 |  |
  G. morbillorum, Eradication: number analyzed (Participants) | 1 | 0 | 0
  G. morbillorum, Eradication | 0 |  |
  G. morbillorum, Presumed eradication: number analyzed (Participants) | 1 | 0 | 0
  G. morbillorum, Presumed eradication | 100 |  |
  G. morbillorum, Persistence: number analyzed (Participants) | 1 | 0 | 0
  G. morbillorum, Persistence | 0 |  |
  G. morbillorum, Presumed persistence: number analyzed (Participants) | 1 | 0 | 0
  G. morbillorum, Presumed persistence | 0 |  |
  G. morbillorum, Indeterminate: number analyzed (Participants) | 1 | 0 | 0
  G. morbillorum, Indeterminate | 0 |  |
  L. lactis, Eradication: number analyzed (Participants) | 1 | 0 | 0
  L. lactis, Eradication | 0 |  |
  L. lactis, Presumed eradication: number analyzed (Participants) | 1 | 0 | 0
  L. lactis, Presumed eradication | 100 |  |
  L. lactis, Persistence: number analyzed (Participants) | 1 | 0 | 0
  L. lactis, Persistence | 0 |  |
  L. lactis, Presumed persistence: number analyzed (Participants) | 1 | 0 | 0
  L. lactis, Presumed persistence | 0 |  |
  L. lactis, Indeterminate: number analyzed (Participants) | 1 | 0 | 0
  L. lactis, Indeterminate | 0 |  |

25. Secondary Outcome: Microbiological Response at the End of Treatment (EOT) Visit by Baseline Gram-positive Pathogen
Description: as for outcome 21
Time Frame: Baseline, Day 14 (± 2 Days)
Population: Participants in the microITT population with specified baseline pathogen
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 52 | 55 | 18
percentage of participants
  S. aureus (MRSA), Eradication: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA), Eradication | 0 | 0 |
  S. aureus (MRSA), Presumed eradication: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA), Presumed eradication | 100 | 75 |
  S. aureus (MRSA), Persistence: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA), Persistence | 0 | 0 |
  S. aureus (MRSA), Presumed persistence: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA), Presumed persistence | 0 | 25 |
  S. aureus (MRSA), Indeterminate: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA), Indeterminate | 0 | 0 |
  S. aureus (MSSA), Eradication: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Eradication | 0 | 2.3 | 0
  S. aureus (MSSA), Presumed eradication: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Presumed eradication | 95.7 | 88.6 | 100
  S. aureus (MSSA), Persistence: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Persistence | 0 | 2.3 | 0
  S. aureus (MSSA), Presumed persistence: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Presumed persistence | 2.1 | 2.3 | 0
  S. aureus (MSSA), Indeterminate: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Indeterminate | 2.1 | 2.3 | 0
  S. aureus (MSSA), Missing: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Missing | 0 | 2.3 | 0
  S. agalactiae, Eradication: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Eradication |  | 0 |
  S. agalactiae, Presumed eradication: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Presumed eradication |  | 100 |
  S. agalactiae, Persistence: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Persistence |  | 0 |
  S. agalactiae, Presumed persistence: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Presumed persistence |  | 0 |
  S. agalactiae, Indeterminate: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Indeterminate |  | 0 |
  S. anginosus, Eradication: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Eradication | 0 |  |
  S. anginosus, Presumed eradication: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Presumed eradication | 100 |  |
  S. anginosus, Persistence: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Persistence | 0 |  |
  S. anginosus, Presumed persistence: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Presumed persistence | 0 |  |
  S. anginosus, Indeterminate: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Indeterminate | 0 |  |
  S. constellatus, Eradication: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Eradication |  | 0 |
  S. constellatus, Presumed eradication: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Presumed eradication |  | 100 |
  S. constellatus, Persistence: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Persistence |  | 0 |
  S. constellatus, Presumed persistence: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Presumed persistence |  | 0 |
  S. constellatus, Indeterminate: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Indeterminate |  | 0 |
  S. intermedius, Eradication: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Eradication |  | 0 |
  S. intermedius, Presumed eradication: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Presumed eradication |  | 100 |
  S. intermedius, Persistence: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Persistence |  | 0 |
  S. intermedius, Presumed persistence: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Presumed persistence |  | 0 |
  S. intermedius, Indeterminate: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Indeterminate |  | 0 |
  S. mitis/oralis, Eradication: number analyzed (Participants) | 1 | 1 | 1
  S. mitis/oralis, Eradication | 0 | 0 | 0
  S. mitis/oralis, Presumed eradication: number analyzed (Participants) | 1 | 1 | 1
  S. mitis/oralis, Presumed eradication | 100 | 100 | 100
  S. mitis/oralis, Persistence: number analyzed (Participants) | 1 | 1 | 1
  S. mitis/oralis, Persistence | 0 | 0 | 0
  S. mitis/oralis, Presumed persistence: number analyzed (Participants) | 1 | 1 | 1
  S. mitis/oralis, Presumed persistence | 0 | 0 | 0
  S. mitis/oralis, Indeterminate: number analyzed (Participants) | 1 | 1 | 1
  S. mitis/oralis, Indeterminate | 0 | 0 | 0
  S. pyogenes, Eradication: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Eradication | 0 | 0 | 0
  S. pyogenes, Presumed eradication: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Presumed eradication | 80 | 75 | 100
  S. pyogenes, Persistence: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Persistence | 0 | 0 | 0
  S. pyogenes, Presumed persistence: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Presumed persistence | 20 | 0 | 0
  S. pyogenes, Indeterminate: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Indeterminate | 0 | 0 | 0
  S. pyogenes, Missing: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Missing | 0 | 25 | 0
  E. faecalis, Eradication: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Eradication | 0 | 0 |
  E. faecalis, Presumed eradication: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Presumed eradication | 100 | 100 |
  E. faecalis, Persistence: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Persistence | 0 | 0 |
  E. faecalis, Presumed persistence: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Presumed persistence | 0 | 0 |
  E. faecalis, Indeterminate: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Indeterminate | 0 | 0 |
  E. hirae, Eradication: number analyzed (Participants) | 1 | 0 | 0
  E. hirae, Eradication | 0 |  |
  E. hirae, Presumed eradication: number analyzed (Participants) | 1 | 0 | 0
  E. hirae, Presumed eradication | 0 |  |
  E. hirae, Persistence: number analyzed (Participants) | 1 | 0 | 0
  E. hirae, Persistence | 0 |  |
  E. hirae, Presumed persistence: number analyzed (Participants) | 1 | 0 | 0
  E. hirae, Presumed persistence | 0 |  |
  E. hirae, Indeterminate: number analyzed (Participants) | 1 | 0 | 0
  E. hirae, Indeterminate | 100 |  |
  G. morbillorum, Eradication: number analyzed (Participants) | 1 | 0 | 0
  G. morbillorum, Eradication | 0 |  |
  G. morbillorum, Presumed eradication: number analyzed (Participants) | 1 | 0 | 0
  G. morbillorum, Presumed eradication | 100 |  |
  G. morbillorum, Persistence: number analyzed (Participants) | 1 | 0 | 0
  G. morbillorum, Persistence | 0 |  |
  G. morbillorum, Presumed persistence: number analyzed (Participants) | 1 | 0 | 0
  G. morbillorum, Presumed persistence | 0 |  |
  G. morbillorum, Indeterminate: number analyzed (Participants) | 1 | 0 | 0
  G. morbillorum, Indeterminate | 0 |  |
  L. lactis, Eradication: number analyzed (Participants) | 1 | 0 | 0
  L. lactis, Eradication | 0 |  |
  L. lactis, Presumed eradication: number analyzed (Participants) | 1 | 0 | 0
  L. lactis, Presumed eradication | 100 |  |
  L. lactis, Persistence: number analyzed (Participants) | 1 | 0 | 0
  L. lactis, Persistence | 0 |  |
  L. lactis, Presumed persistence: number analyzed (Participants) | 1 | 0 | 0
  L. lactis, Presumed persistence | 0 |  |
  L. lactis, Indeterminate: number analyzed (Participants) | 1 | 0 | 0
  L. lactis, Indeterminate | 0 |  |

26. Secondary Outcome: Microbiological Response at the Test of Cure (TOC) Visit by Baseline Gram-positive Pathogen
Description: as for outcome 22
Time Frame: Baseline, Day 28 (± 2 Days)
Population: Participants in the microITT population with specified baseline pathogen
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 52 | 55 | 18
percentage of participants
  S. aureus (MRSA), Eradication: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA), Eradication | 0 | 0 |
  S. aureus (MRSA), Presumed eradication: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA), Presumed eradication | 100 | 75 |
  S. aureus (MRSA), Persistence: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA), Persistence | 0 | 0 |
  S. aureus (MRSA), Presumed persistence: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA), Presumed persistence | 0 | 25 |
  S. aureus (MRSA), Indeterminate: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA), Indeterminate | 0 | 0 |
  S. aureus (MSSA), Eradication: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Eradication | 0 | 2.3 | 0
  S. aureus (MSSA), Presumed eradication: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Presumed eradication | 91.5 | 88.6 | 100
  S. aureus (MSSA), Persistence: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Persistence | 0 | 0 | 0
  S. aureus (MSSA), Presumed persistence: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Presumed persistence | 2.1 | 4.5 | 0
  S. aureus (MSSA), Indeterminate: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Indeterminate | 6.4 | 2.3 | 0
  S. aureus (MSSA), Missing: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Missing | 0 | 2.3 | 0
  S. agalactiae, Eradication: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Eradication |  | 0 |
  S. agalactiae, Presumed eradication: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Presumed eradication |  | 100 |
  S. agalactiae, Persistence: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Persistence |  | 0 |
  S. agalactiae, Presumed persistence: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Presumed persistence |  | 0 |
  S. agalactiae, Indeterminate: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Indeterminate |  | 0 |
  S. anginosus, Eradication: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Eradication | 0 |  |
  S. anginosus, Presumed eradication: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Presumed eradication | 100 |  |
  S. anginosus, Persistence: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Persistence | 0 |  |
  S. anginosus, Presumed persistence: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Presumed persistence | 0 |  |
  S. anginosus, Indeterminate: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Indeterminate | 0 |  |
  S. constellatus, Eradication: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Eradication |  | 0 |
  S. constellatus, Presumed eradication: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Presumed eradication |  | 100 |
  S. constellatus, Persistence: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Persistence |  | 0 |
  S. constellatus, Presumed persistence: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Presumed persistence |  | 0 |
  S. constellatus, Indeterminate: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Indeterminate |  | 0 |
  S. intermedius, Eradication: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Eradication |  | 0 |
  S. intermedius, Presumed eradication: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Presumed eradication |  | 100 |
  S. intermedius, Persistence: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Persistence |  | 0 |
  S. intermedius, Presumed persistence: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Presumed persistence |  | 0 |
  S. intermedius, Indeterminate: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Indeterminate |  | 0 |
  S. mitis/oralis, Eradication: number analyzed (Participants) | 1 | 1 | 1
  S. mitis/oralis, Eradication | 0 | 0 | 0
  S. mitis/oralis, Presumed eradication: number analyzed (Participants) | 1 | 1 | 1
  S. mitis/oralis, Presumed eradication | 100 | 100 | 100
  S. mitis/oralis, Persistence: number analyzed (Participants) | 1 | 1 | 1
  S. mitis/oralis, Persistence | 0 | 0 | 0
  S. mitis/oralis, Presumed persistence: number analyzed (Participants) | 1 | 1 | 1
  S. mitis/oralis, Presumed persistence | 0 | 0 | 0
  S. mitis/oralis, Indeterminate: number analyzed (Participants) | 1 | 1 | 1
  S. mitis/oralis, Indeterminate | 0 | 0 | 0
  S. pyogenes, Eradication: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Eradication | 0 | 0 | 0
  S. pyogenes, Presumed eradication: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Presumed eradication | 80 | 75 | 100
  S. pyogenes, Persistence: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Persistence | 0 | 0 | 0
  S. pyogenes, Presumed persistence: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Presumed persistence | 20 | 0 | 0
  S. pyogenes, Indeterminate: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Indeterminate | 0 | 0 | 0
  S. pyogenes, Missing: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Missing | 0 | 25 | 0
  E. faecalis, Eradication: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Eradication | 0 | 0 |
  E. faecalis, Presumed eradication: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Presumed eradication | 100 | 100 |
  E. faecalis, Persistence: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Persistence | 0 | 0 |
  E. faecalis, Presumed persistence: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Presumed persistence | 0 | 0 |
  E. faecalis, Indeterminate: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Indeterminate | 0 | 0 |
  E. hirae, Eradication: number analyzed (Participants) | 1 | 0 | 0
  E. hirae, Eradication | 0 |  |
  E. hirae, Presumed eradication: number analyzed (Participants) | 1 | 0 | 0
  E. hirae, Presumed eradication | 100 |  |
  E. hirae, Persistence: number analyzed (Participants) | 1 | 0 | 0
  E. hirae, Persistence | 0 |  |
  E. hirae, Presumed persistence: number analyzed (Participants) | 1 | 0 | 0
  E. hirae, Presumed persistence | 0 |  |
  E. hirae, Indeterminate: number analyzed (Participants) | 1 | 0 | 0
  E. hirae, Indeterminate | 0 |  |
  G. morbillorum, Eradication: number analyzed (Participants) | 1 | 0 | 0
  G. morbillorum, Eradication | 0 |  |
  G. morbillorum, Presumed eradication: number analyzed (Participants) | 1 | 0 | 0
  G. morbillorum, Presumed eradication | 100 |  |
  G. morbillorum, Persistence: number analyzed (Participants) | 1 | 0 | 0
  G. morbillorum, Persistence | 0 |  |
  G. morbillorum, Presumed persistence: number analyzed (Participants) | 1 | 0 | 0
  G. morbillorum, Presumed persistence | 0 |  |
  G. morbillorum, Indeterminate: number analyzed (Participants) | 1 | 0 | 0
  G. morbillorum, Indeterminate | 0 |  |
  L. lactis, Eradication: number analyzed (Participants) | 1 | 0 | 0
  L. lactis, Eradication | 0 |  |
  L. lactis, Presumed eradication: number analyzed (Participants) | 1 | 0 | 0
  L. lactis, Presumed eradication | 100 |  |
  L. lactis, Persistence: number analyzed (Participants) | 1 | 0 | 0
  L. lactis, Persistence | 0 |  |
  L. lactis, Presumed persistence: number analyzed (Participants) | 1 | 0 | 0
  L. lactis, Presumed persistence | 0 |  |
  L. lactis, Indeterminate: number analyzed (Participants) | 1 | 0 | 0
  L. lactis, Indeterminate | 0 |  |

27. Secondary Outcome: Microbiological Response at the Follow-Up Visit by Baseline Gram-positive Pathogen
Description: as for outcome 22
Time Frame: Baseline, Day 54 (± 7 days)
Population: Participants in the microITT population with specified baseline pathogen
Measure: Number; unit: percentage of participants
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
Number analyzed (Participants) | 52 | 55 | 18
percentage of participants
  S. aureus (MRSA), Eradication: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA), Eradication | 0 | 0 |
  S. aureus (MRSA), Presumed eradication: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA), Presumed eradication | 50 | 50 |
  S. aureus (MRSA), Persistence: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA), Persistence | 0 | 0 |
  S. aureus (MRSA), Presumed persistence: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA), Presumed persistence | 0 | 25 |
  S. aureus (MRSA), Indeterminate: number analyzed (Participants) | 2 | 4 | 0
  S. aureus (MRSA), Indeterminate | 50 | 25 |
  S. aureus (MSSA), Eradication: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Eradication | 0 | 2.3 | 0
  S. aureus (MSSA), Presumed eradication: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Presumed eradication | 93.6 | 86.4 | 100
  S. aureus (MSSA), Persistence: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Persistence | 0 | 0 | 0
  S. aureus (MSSA), Presumed persistence: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Presumed persistence | 2.1 | 4.5 | 0
  S. aureus (MSSA), Indeterminate: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Indeterminate | 4.3 | 4.5 | 0
  S. aureus (MSSA), Missing: number analyzed (Participants) | 47 | 44 | 14
  S. aureus (MSSA), Missing | 0 | 2.3 | 0
  S. agalactiae, Eradication: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Eradication |  | 0 |
  S. agalactiae, Presumed eradication: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Presumed eradication |  | 100 |
  S. agalactiae, Persistence: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Persistence |  | 0 |
  S. agalactiae, Presumed persistence: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Presumed persistence |  | 0 |
  S. agalactiae, Indeterminate: number analyzed (Participants) | 0 | 1 | 0
  S. agalactiae, Indeterminate |  | 0 |
  S. anginosus, Eradication: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Eradication | 0 |  |
  S. anginosus, Presumed eradication: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Presumed eradication | 100 |  |
  S. anginosus, Persistence: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Persistence | 0 |  |
  S. anginosus, Presumed persistence: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Presumed persistence | 0 |  |
  S. anginosus, Indeterminate: number analyzed (Participants) | 1 | 0 | 0
  S. anginosus, Indeterminate | 0 |  |
  S. constellatus, Eradication: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Eradication |  | 0 |
  S. constellatus, Presumed eradication: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Presumed eradication |  | 100 |
  S. constellatus, Persistence: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Persistence |  | 0 |
  S. constellatus, Presumed persistence: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Presumed persistence |  | 0 |
  S. constellatus, Indeterminate: number analyzed (Participants) | 0 | 1 | 0
  S. constellatus, Indeterminate |  | 0 |
  S. intermedius, Eradication: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Eradication |  | 0 |
  S. intermedius, Presumed eradication: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Presumed eradication |  | 100 |
  S. intermedius, Persistence: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Persistence |  | 0 |
  S. intermedius, Presumed persistence: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Presumed persistence |  | 0 |
  S. intermedius, Indeterminate: number analyzed (Participants) | 0 | 1 | 0
  S. intermedius, Indeterminate |  | 0 |
  S. mitis/oralis, Eradication: number analyzed (Participants) | 1 | 1 | 1
  S. mitis/oralis, Eradication | 0 | 0 | 0
  S. mitis/oralis, Presumed eradication: number analyzed (Participants) | 1 | 1 | 1
  S. mitis/oralis, Presumed eradication | 100 | 100 | 100
  S. mitis/oralis, Persistence: number analyzed (Participants) | 1 | 1 | 1
  S. mitis/oralis, Persistence | 0 | 0 | 0
  S. mitis/oralis, Presumed persistence: number analyzed (Participants) | 1 | 1 | 1
  S. mitis/oralis, Presumed persistence | 0 | 0 | 0
  S. mitis/oralis, Indeterminate: number analyzed (Participants) | 1 | 1 | 1
  S. mitis/oralis, Indeterminate | 0 | 0 | 0
  S. pyogenes, Eradication: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Eradication | 0 | 0 | 0
  S. pyogenes, Presumed eradication: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Presumed eradication | 80 | 75 | 100
  S. pyogenes, Persistence: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Persistence | 0 | 0 | 0
  S. pyogenes, Presumed persistence: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Presumed persistence | 20 | 0 | 0
  S. pyogenes, Indeterminate: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Indeterminate | 0 | 0 | 0
  S. pyogenes, Missing: number analyzed (Participants) | 5 | 4 | 3
  S. pyogenes, Missing | 0 | 25 | 0
  E. faecalis, Eradication: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Eradication | 0 | 0 |
  E. faecalis, Presumed eradication: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Presumed eradication | 100 | 100 |
  E. faecalis, Persistence: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Persistence | 0 | 0 |
  E. faecalis, Presumed persistence: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Presumed persistence | 0 | 0 |
  E. faecalis, Indeterminate: number analyzed (Participants) | 2 | 2 | 0
  E. faecalis, Indeterminate | 0 | 0 |
  E. hirae, Eradication: number analyzed (Participants) | 1 | 0 | 0
  E. hirae, Eradication | 0 |  |
  E. hirae, Presumed eradication: number analyzed (Participants) | 1 | 0 | 0
  E. hirae, Presumed eradication | 100 |  |
  E. hirae, Persistence: number analyzed (Participants) | 1 | 0 | 0
  E. hirae, Persistence | 0 |  |
  E. hirae, Presumed persistence: number analyzed (Participants) | 1 | 0 | 0
  E. hirae, Presumed persistence | 0 |  |
  E. hirae, Indeterminate: number analyzed (Participants) | 1 | 0 | 0
  E. hirae, Indeterminate | 0 |  |
  G. morbillorum, Eradication: number analyzed (Participants) | 1 | 0 | 0
  G. morbillorum, Eradication | 0 |  |
  G. morbillorum, Presumed eradication: number analyzed (Participants) | 1 | 0 | 0
  G. morbillorum, Presumed eradication | 100 |  |
  G. morbillorum, Persistence: number analyzed (Participants) | 1 | 0 | 0
  G. morbillorum, Persistence | 0 |  |
  G. morbillorum, Presumed persistence: number analyzed (Participants) | 1 | 0 | 0
  G. morbillorum, Presumed persistence | 0 |  |
  G. morbillorum, Indeterminate: number analyzed (Participants) | 1 | 0 | 0
  G. morbillorum, Indeterminate | 0 |  |
  L. lactis, Eradication: number analyzed (Participants) | 1 | 0 | 0
  L. lactis, Eradication | 0 |  |
  L. lactis, Presumed eradication: number analyzed (Participants) | 1 | 0 | 0
  L. lactis, Presumed eradication | 100 |  |
  L. lactis, Persistence: number analyzed (Participants) | 1 | 0 | 0
  L. lactis, Persistence | 0 |  |
  L. lactis, Presumed persistence: number analyzed (Participants) | 1 | 0 | 0
  L. lactis, Presumed persistence | 0 |  |
  L. lactis, Indeterminate: number analyzed (Participants) | 1 | 0 | 0
  L. lactis, Indeterminate | 0 |  |

28. Secondary Outcome: All-cause Mortality at the Test of Cure (TOC) Visit Among Cohort 5 Participants
Description: All-cause mortality was determined for the participants in Cohort 5 (birth to < 3 months) at the Test of Cure visit.
Time Frame: Day 28 (± 2 Days)
Population: All participants in the ITT population
Measure: Count of Participants; unit: Participants
Groups:
- Birth to < 3 Months of Age (Cohort 5): Participants aged birth to < 3 months
Arm/Group | Birth to < 3 Months of Age (Cohort 5)
Number analyzed (Participants) | 10
Participants | 0

29. Secondary Outcome: Concentration of Dalbavancin in Plasma
Description: The population pharmacokinetic (PK) profile of dalbavancin was assessed using a sparse sampling approach. Plasma PK samples were collected from participants receiving dalbavancin treatment (single-dose and two-dose arms) at 30 minutes and at 2 hours (Day 1), at 48-72 hours (Day 3-4), at 168 ± 24 hours (Day 8 ± 1), and at 312 ± 48 hours and analyzed for dalbavancin concentration.
Time Frame: 30 min (end of infusion on Day 1); 2 hrs after start of IV (Day 1); and 48-72 hrs, 168 hrs, and 312 hrs after start of IV
Population: All participants in the ITT population who received at least 1 dose of study drug with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- 3 Months to < 2 Years Old (Cohort 4): Participants aged 3 months to < 2 years old
- 2 Years to < 6 Years Old (Cohort 3): Participants aged 2 years to < 6 years old
- Participants Aged 6 Years to < 12 Years Old: Participants aged 6 years to < 12 years old
- 12 Years to 17 Years Old (Cohort 1): Participants aged 12 years to 17 years old
Arm/Group | Birth to < 3 Months of Age (Cohort 5) | 3 Months to < 2 Years Old (Cohort 4) | 2 Years to < 6 Years Old (Cohort 3) | Participants Aged 6 Years to < 12 Years Old | 12 Years to 17 Years Old (Cohort 1)
Number analyzed (Participants) | 10 | 16 | 34 | 49 | 58
µg/mL
  30 min (end of infusion): number analyzed (Participants) | 10 | 15 | 33 | 49 | 58
  30 min (end of infusion) | 212.43 (23.32) | 268.02 (44.90) | 219.45 (66.72) | 211.30 (34.26) | 233.58 (46.44)
  2 hrs after start of IV: number analyzed (Participants) | 10 | 15 | 34 | 49 | 58
  2 hrs after start of IV | 133.83 (24.66) | 196.51 (53.44) | 149.28 (43.40) | 165.75 (37.46) | 162.54 (36.85)
  48-72 hrs after start of IV: number analyzed (Participants) | 10 | 16 | 33 | 49 | 57
  48-72 hrs after start of IV | 53.53 (24.48) | 61.32 (40.08) | 56.68 (46.25) | 56.93 (39.79) | 60.92 (28.68)
  168 hrs after start of IV: number analyzed (Participants) | 10 | 13 | 31 | 49 | 57
  168 hrs after start of IV | 16.89 (35.12) | 28.80 (119.04) | 24.10 (80.90) | 26.25 (51.38) | 31.41 (31.24)
  312 hrs after start of IV: number analyzed (Participants) | 10 | 12 | 30 | 47 | 56
  312 hrs after start of IV | 4.94 (47.91) | 15.24 (47.97) | 12.74 (45.62) | 15.35 (39.40) | 20.75 (37.71)

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse events were collected from the time informed consent was signed through the Final Visit. Median time on follow-up was 54.0 days for the Dalbavancin Single-dose and Dalbavancin Two-dose groups and 54.5 days for the Comparator group.
Description: Adverse events were analyzed in the safety population which is defined as all participants in the ITT population who received at least 1 dose of study drug.
Arm/Group | Dalbavancin Single-dose | Dalbavancin Two-dose | Comparator
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/78 | 0/30
Serious Adverse Events (participants affected / at risk) | 3/91 | 0/78 | 0/30
Other Adverse Events (participants affected / at risk) | 1/91 | 5/78 | 1/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalbavancin Single-dose (N=91) | Dalbavancin Two-dose (N=78) | Comparator (N=30)
ABSCESS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OSTEOMYELITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
FEBRILE CONVULSION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalbavancin Single-dose (N=91) | Dalbavancin Two-dose (N=78) | Comparator (N=30)
VOMITING (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 2 (2) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT02814916/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/16/NCT02814916/SAP_001.pdf